CLINICAL TRIAL: NCT02595008
Title: An Open Label, Safety Study to Assess the Potential for Adrenal Suppression and Pharmacokinetics Following Maximal Use Treatment With DSXS in Patients With Atopic Dermatitis.
Brief Title: Study to Assess the Potential for Adrenal Suppression Following Treatment With DSXS in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSXS 1502
Record Dates: First submitted 2015-11-01; First posted 2015-11-03 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DSXS topical product (Experimental): treatment with DSXS twice daily for 28 days
  Interventions: Drug: DSXS

INTERVENTIONS:
Drug: DSXS — Active treatment
  Other Names: Active

SUMMARY:
this study is to evaluate the potential of DSXS to suppress HPA axis function in patients with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the potential of DSXS to suppress HPA axis function in patients with moderate to severe atopic dermatitis.

The secondary objectives are to evaluate to evaluate adverse event (AE) profiles of DSXS administered to patients with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a definite clinical diagnosis of stable atopic dermatitis

Exclusion Criteria:

* Patient is under the age of 2

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08-28 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novum Pharmaceutical Research Services, Study Chair — http://www.novumprs.com/contact
Locations (1):
- Taro Pharmaceuticals USA Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DSXS Topical Product Cohort 1: treatment with DSXS twice daily for 28 days in patients age 18 years and older
  DSXS: Active treatment
- DSXS Topical Product Cohort 2: treatment with DSXS twice daily for 28 days in patients age 12-17 years of age
  DSXS: Active treatment
Period: Overall Study
Arm/Group | DSXS Topical Product Cohort 1 | DSXS Topical Product Cohort 2
Started | 20 | 4
Completed | 19 | 4
Not Completed | 1 | 0
Not completed — Enrolled In Error | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DSXS Topical Product Cohort 1 | DSXS Topical Product Cohort 2 | Total
Number analyzed (Participants) | 19 | 4 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.32 (11.18) | 15.25 (2.36) | 38.43 (14.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 12
  Male | 9 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 2 | 15
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 14 | 3 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Total BSA [Mean (Standard Deviation); unit: meters squared] | 2.03 (0.29) | 1.78 (0.31) | 1.98 (0.30)
Baseline IGA [Count of Participants; unit: Participants]
  Clear | 0 | 0 | 0
  Almost Clear | 0 | 0 | 0
  Mild Disease | 0 | 0 | 0
  Moderate Disease | 17 | 2 | 19
  Severe Disease | 2 | 2 | 4
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: units on a scale] — The EASI is a composite score based on the severity of four different signs of atopic dermatitis (Erythema, Induration/Papulation/Edema, Lichenification, and Excoriation rated 0 to 3 in severity) in four different areas of the body (Head/Neck, Upper Limbs, Trunk, Lower Limbs) multiplied by the percent of that specific body area affected multiplied by a weighting factor. The minimum score would be 0 and the maximum score would be 72. To be eligible for participation in this study a patient must have an EASI of at least 15 at baseline. A higher EASI value represents a more severe case of eczema.
  units on a scale | 19.74 (9.08) | 28.50 (19.91) | 21.26 (11.53)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HPA Axis Suppression
Description: Hypothalamic Pituitary Adrenal (HPA) Axis Response to Cosyntropin demonstrating the absence or presence of adrenal suppression at the end of treatment. HPA Axis suppression is defined as a 30 minute post CortrosynTM injection level cortisol level of ≤ 18 mcg/100ml.
Time Frame: 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS Topical Product Cohort 1 | DSXS Topical Product Cohort 2
Number analyzed (Participants) | 19 | 4
Participants
  Yes | 3 | 1
  No | 16 | 3

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Arm/Group | DSXS Topical Product Cohort 1 | DSXS Topical Product Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/4
Other Adverse Events (participants affected / at risk) | 4/19 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSXS Topical Product Cohort 1 (N=19) | DSXS Topical Product Cohort 2 (N=4)
ACTH stimulation test abnormal (Investigations) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-09-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT02595008/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT02595008/SAP_001.pdf